CLINICAL TRIAL: NCT02609503
Title: Pembrolizumab and Radiation for Locally Advanced Squamous Cell Carcinoma of the Head and Neck (SCCHN) Not Eligible for Cisplatin Therapy
Brief Title: Pembrolizumab + Radiation for Locally Adv SCC of the Head and Neck (SCCHN) Not Eligible Cisplatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1509
Record Dates: First submitted 2015-11-12; First posted 2015-11-20 (Estimated); Results first posted 2021-03-19 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — pembrolizumab; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open label (Experimental): Pembrolizumab
  Interventions: Drug: Pembrolizumab
- Radiation (Other): Intensity Modulated Radiation Therapy (IMRT)
  Interventions: Radiation: Intensity Modulated Radiation Therapy

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab, 200 mg IV during cycle visits every 3-weeks for up to 6 cycles, or until toxicities are no longer tolerable
  Other Names: Keytruda
  Arms: Open label
Radiation: Intensity Modulated Radiation Therapy — Eligible participants will receive Intensity Modulated Radiation Therapy daily x 7 weeks
  Other Names: IMRT
  Arms: Radiation

SUMMARY:
This study is being done to evaluate the efficacy of Pembrolizumab, concomitant with and following standard of care definitive radiation, for locally advanced squamous cell carcinoma of the head and neck patients who are not good candidates for Cisplatin.

DETAILED DESCRIPTION:
This open label, phase II trial will enroll 29 subjects in order to evaluate the efficacy of Pembrolizumab, concomitant with and following standard of care definitive radiation for locally advanced squamous cell carcinoma head and neck patients who are not good candidates for Cisplatin. Objectives include estimating progression free survival and overall survival, response rates, safety and toxicity, and quality of life in these patients. Correlative studies, based on serial blood collections and tumor samples, may be done under a separate protocol based on availability of archival diagnostic tissue.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial
* Be greater than or equal to 18 years of age
* Eastern Cooperative Oncology Group (ECOG) Performance Status less than or equal to 1
* Histologically or cytologically confirmed stage III-IV (non-metastatic) squamous cell carcinoma of the head and neck as defined by American Joint Committee on Cancer. Nasopharyngeal cancer patients will be excluded.
* Ineligible for high dose cisplatin therapy; the reason for ineligibility must be defined.
* Demonstrate adequate organ function. All screening labs should be performed within 14 days of treatment initiation.
* No prior curative attempts for this cancer (i.e., surgery, radiation and/or other).
* Female patients of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. Serum pregnancy test may be required.
* Female patients of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication.
* Male patients should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* As determined by the enrolling physician or protocol designee, ability of the patient to understand and comply with study procedures for the entire length of the study.
* Consent for the use of any residual material from biopsy (archival tissue) and serial blood draws will be required for enrollment.

Exclusion Criteria:

* If currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered from adverse events due to agents administered more than 4 weeks earlier
* Had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered from adverse events due to a previously administered agent.
* Has a known additional malignancy that is metastatic, progressing or requires active treatment.
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease even if resolved; patients with vitiligo or resolved childhood asthma/atopy would be an exception to this rule.
* Has clinical or radiologic evidence of interstitial lung disease or active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Has inadequate home environment or social support to safely complete the trial procedures.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-programmed cell death (PD-1), anti-PD-L1, anti-PD-L1, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody.
* Has a known history of Human Immunodeficiency Virus (HIV) HIV 1/2 antibodies) Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C )e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2023-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Weiss, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (3):
- United States (3):
  - John Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Weiss J, Sheth S, Deal AM, Grilley Olson JE, Patel S, Hackman TG, Blumberg JM, Galloway TJ, Patel S, Zanation AM, Shen CJ, Hayes DN, Hilliard C, Mehra R, McKinnon KP, Wang HH, Weissler MC, Bauman JR, Chera BS, Vincent BG. Concurrent Definitive Immunoradiotherapy for Patients with Stage III-IV Head and Neck Cancer and Cisplatin Contraindication. Clin Cancer Res. 2020 Aug 15;26(16):4260-4267. doi: 10.1158/1078-0432.CCR-20-0230. Epub 2020 May 5. PMID 32371539
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the University of North Carolina (Chapel Hill, NC), Fox Chase Cancer Center (Philadelphia, PA), and Johns Hopkins (Baltimore,MD) between February 2016 and July 2018.
Pre-assignment Details: One potential participant was deemed ineligible during screening and therefore did not start the trial.
Groups:
- Pembrolizumab Concomitant With and Post 7 Weeks of Radiation: All patients will receive Intensity Modulated Radiotherapy Treatments (IMRT) as per standard of care. The total dose will be 70 Gray(Gy) at 2Gy/fraction, 35 fractions, Monday to Friday, for 7 weeks.
  Starting on the first day of radiotherapy, patients will be treated with pembrolizumab 200 milligrams (mg) intravenous (IV) every 3 weeks for 6 doses.
Period: Overall Study
Arm/Group | Pembrolizumab Concomitant With and Post 7 Weeks of Radiation
Started | 29
Completed | 25
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Disease progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab Concomitant With and Post 7 Weeks of Radiation
Number analyzed (Participants) | 29
Age, Continuous [Mean (Full Range); unit: years] | 63.1 [39 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 29
Smoking status [Count of Participants; unit: Participants]
  Current | 3
  Former | 15
  Never | 11
Smoking pack years [Count of Participants; unit: Participants] — For former/current smokers, an estimate of how much they have smoked.
  Participants
    <10 pack years | 13
    >=10 pack years | 16
Performance status [Count of Participants; unit: Participants] — East Coast Oncology Group (ECOG) Performance status: 0-5 scale to describe a patient's level of functioning in terms of selfcare ability and activity level (lower score means higher functioning) 0-Fully active
  1. Restricted in strenuous activity but ambulatory and able to carry out light work
  2. Ambulatory, capable of all selfcare but unable to carry out any work; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; can't carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 12
    1 | 17
Reason for cisplatin ineligibility [Count of Participants; unit: Participants]
  Hearing | 14
  Tinnitus | 6
  Renal function | 5
  Diabetes | 2
  Neuropathy | 2
Charleson comorbidity index score [Count of Participants; unit: Participants] — The Charlson Comorbidity Index is a method of categorizing comorbidities of patients in which each category has an associated weight (from 1 to 6), based on the adjusted risk of mortality or resource use, and the sum of all the weights results in a single comorbidity score for a patient ranging from 0 (no comorbidities) to 24. The higher the score, the more likely the predicted outcome will result in mortality or higher resource use.
  Participants
    0 | 6
    1 | 6
    2 | 11
    3 | 2
    4 | 3
    5 | 1
Primary site [Count of Participants; unit: Participants]
  Base of tongue | 10
  Tonsil | 10
  Supraglottic larynx | 3
  Hypopharynx | 2
  Unknown primary | 2
  Oral tongue | 1
  Uvula | 1
Stage [Count of Participants; unit: Participants] — Anatomic stage is the American Joint Committee on Cancer (AJCC) system, which is based on:
  Size of primary tumor (T) and whether it has grown into nearby areas. Spread to regional lymph nodes (N). Spread (metastasis; M) to other organs of the body. Once the T, N, and M categories have been determined, this information is combined into a prognostic stage group. Higher Roman numerals mean the cancer is more advanced.
  Participants
    I | 5
    II | 3
    III | 11
    IVA | 8
    IVB | 2
Programmed cell Death Ligand-1 (PD-L1) Modified Percent Score (MPS) [Median (Full Range); unit: percent staining] — The percent of tumor with membrane-specific staining was directly estimated at four intensity levels [negative (<1), low (1+), moderate (2+), and high (3+)] and reported as a percentage quantitatively as any one of the following: 0%, 1%, 2%, 5%, 10%, 15%, 20%, 30%, 40%, 50%, 60%, 70%, 80%, 85%, 90%, 93%, 95%, 99%, or 100%. To calculate MPS, the percents of tumor staining at low, moderate, and high levels were summed. The potential range of the scale is from 0 to 100 with a higher score indicating higher PD-L1.
  percent staining | 60 [0 to 100]
Programmed cell Death Ligand-1 (PD-L1) modified H-score (MHS) [Median (Full Range); unit: units on a scale] — The percent of tumor with membrane-specific staining was directly estimated at four intensity levels [negative (<1), low (1+), moderate (2+), and high (3+)] and reported as a percentage quantitatively. To calculate MHS, the percent of membrane staining at low levels was multiplied by a factor of 1, the percent of staining at moderate levels was multiplied by 2, and the percent of staining at high levels was multiplied by 3; the three products were then summed to arrive at a final MHS. Potential range of scale is 0 to 300, with a higher score indicating higher expression of PD-L1.
  units on a scale | 105 [0 to 280]
Tumor-Infiltrating Lymphocytes (TIL) [Median (Full Range); unit: units on a scale] — The abundance of TILs present was noted as a number between 0-3 with 0 being the absence of TILs and 3 indicating high profusion of TILs.
  units on a scale | 3 [0 to 3]

OUTCOME MEASURES:

1. Primary Outcome: 20 Week Progression Free Survival Rate
Description: the proportion of patients who are alive and free of progression from disease at 20 weeks from the start of treatment
Time Frame: 20 weeks after D1 of treatment
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Pembrolizumab Concomitant With and Post 7 Weeks of Radiation
Number analyzed (Participants) | 29
proportion of participants | 0.90 [0.71 to 0.96]

2. Primary Outcome: One Year Progression Free Survival Rate
Description: the proportion of patients who are alive and free of progression from disease atoneyears from the start of treatment
Time Frame: 1 years after D1 of treatment
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Pembrolizumab Concomitant With and Post 7 Weeks of Radiation
Number analyzed (Participants) | 29
proportion of participants | 0.76 [0.56 to 0.88]

3. Primary Outcome: Two Year Progression Free Survival Rate
Description: the proportion of patients who are alive and free of progression from disease at two years from the start of treatment
Time Frame: 2 years after D1 of treatment
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Pembrolizumab Concomitant With and Post 7 Weeks of Radiation
Number analyzed (Participants) | 29
proportion of participants | 0.71 [0.49 to 0.84]

4. Primary Outcome: Median Progression Free Survival
Description: Progression-free survival is defined as the time from D1 of treatment to progression or death from any cause. The median was not reached, thus Kaplan Meier's estimated rate at 5 years is reported.
Time Frame: up to 5 years after D1 of treatment
Population: Participants started the study treatment.
Measure: Mean (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Pembrolizumab Concomitant With and Post 7 Weeks of Radiation
Number analyzed (Participants) | 29
Proportion of participants | 58.6 [38.8 to 74.0]

5. Secondary Outcome: One Year Overall Survival Rate
Description: the proportion of patients who are alive at one year after Day 1 of treatment
Time Frame: 1 year after Day 1 of treatment
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Pembrolizumab Concomitant With and Post 7 Weeks of Radiation
Number analyzed (Participants) | 29
proportion of participants | 0.86 [0.67 to 0.95]

6. Secondary Outcome: Two Year Overall Survival Rate
Description: the proportion of patients who are alive at two years after Day 1 of treatment
Time Frame: 2 years after Day 1 of treatment
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Pembrolizumab Concomitant With and Post 7 Weeks of Radiation
Number analyzed (Participants) | 29
proportion of participants | 0.75 [0.51 to 0.88]

7. Secondary Outcome: Proportion of Participants Who Received <95% of Intended Dose of Radiation
Description: Evaluate the safety of the proposed regimen by Estimating the proportion of patients who receive <95% of the intended dose of radiation (i.e., <67 Gray)
Time Frame: 7 weeks
Measure: Number; unit: proportion of participants
Arm/Group | Pembrolizumab Concomitant With and Post 7 Weeks of Radiation
Number analyzed (Participants) | 29
proportion of participants | 0

8. Secondary Outcome: Number of Participants With Clinically Relevant Adverse Events
Description: Safety was assessed by documenting clinically relevant adverse events, defined as events reported by both the clinician and participant related to concurrent radiation plus pembrolizumab. Clinicians classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 4.0). The grading (severity) scale for each AE term: Grade (G) 1 Mild; asymptomatic/mild symptoms; clinical/diagnostic observations only; G 2 Moderate; G 3 Severe or medically significant but not immediately life-threatening; hospitalization/prolongation of hospitalization indicated; disabling; G 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE. Patient assessed toxicity were classified based on the Patient-Reported Outcome version of the CTCAE (PRO-CTCAE) which measures the severity, interference, and frequency of events on a 5 point likert scale (0-4) with a higher score indicating worse or more bothersome event
Time Frame: Monitored continuously from D1 of treatment through 40 weeks.
Measure: Number; unit: participants
Arm/Group | Pembrolizumab Concomitant With and Post 7 Weeks of Radiation
Number analyzed (Participants) | 29
participants
  Pain | 10
  Decreased appetite | 5
  Swallowing difficulty | 12
  Dry mouth | 24
  Fatigue | 18

9. Secondary Outcome: Overall Response Rate
Description: Overall response rate will be determined per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) which defines Complete Response (CR) as Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; and Overall Response Rate (ORR) = CR + PR/total number of subjects.
Time Frame: 2 years after start of treatment
Population: Two participants did not complete follow-up radiographic measurements to assess for response
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab Concomitant With and Post 7 Weeks of Radiation
Number analyzed (Participants) | 27
Participants | 26

10. Secondary Outcome: Complete Response Rate
Description: complete response rate will be determined using RECIST 1.1 and is defined as the percentage of participants who achieve a Complete response (CR)-Disappearance of all target lesions. Any pathological lymph node (LN) (whether target or non-target) must have decreased in short axis to <10mm.
Time Frame: 2 years after start of treatment
Population: Two participants did not complete follow-up radiographic measurements to assess for response
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab Concomitant With and Post 7 Weeks of Radiation
Number analyzed (Participants) | 27
Participants | 23

11. Secondary Outcome: Five Years Locoregional Recurrence Rate
Description: Time to locoregional recurrence is defined from Day 1 of treatment until the first locoregional progression
Time Frame: 5 years from start of treatment
Population: Subjects started to the study treatment.
Measure: Median (95% Confidence Interval); unit: percentage
Arm/Group | Pembrolizumab Concomitant With and Post 7 Weeks of Radiation
Number analyzed (Participants) | 29
percentage | 19.8 [8.5 to 41.2]

12. Secondary Outcome: Five Years Distant Metastasis Rate
Description: Time to distant metastasis is defined as the time from day 1 of treatment to progression of disease at a distant site; deaths or other progressions will be censored
Time Frame: 5 years from start of treatment
Measure: Median (95% Confidence Interval); unit: percentage
Arm/Group | Pembrolizumab Concomitant With and Post 7 Weeks of Radiation
Number analyzed (Participants) | 29
percentage | 3.8 [0.6 to 24.3]

13. Secondary Outcome: Quality of Life Measured by Functional Assessment of Cancer Therapy - Head and Neck (FACT-HN)
Description: The FACT-HN is the FACT-General (FACT-G) and a head and neck cancer specific (HNC) subscale given at baseline, at end of treatment, and at first follow-up visit. The FACT-G is a measure of general QOL with Items rated by patients on a Likert scale from 0 to 4, assessing function in 4 domains: physical well-being (PWB) (7 items, score range 0-28), social-family well-being (SFWB) (7 items, score range 0-28), emotional well-being (EWB) (6 items, score range 0-24) and functional well-being (FWB) (7 items, score range 0-28). The HNC subscale has 12 items and a score range from 0 to 48. Higher scores represent better QOL.
Time Frame: At baseline, 10 and 20 weeks after initiation of treatment
Population: Three subjects did not complete the FACT assessments and are therefore not included
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Baseline Assessment - Pembrolizumab Concomitant With and Post 7 Weeks of Radiation: Baseline Quality of life Measurements
  All patients will receive Intensity Modulated Radiotherapy Treatments (IMRT) as per standard of care. The total dose will be 70 Gray(Gy) at 2Gy/fraction, 35 fractions, Monday to Friday, for 7 weeks.
  Starting on the first day of radiotherapy, patients will be treated with pembrolizumab 200 milligrams (mg) intravenous (IV) every 3 weeks for 6 doses.
- Week 10 Assessment - Pembrolizumab Concomitant With and Post 7 Weeks of Radiation: Week 10 Quality of life Measurements
  All patients will receive Intensity Modulated Radiotherapy Treatments (IMRT) as per standard of care. The total dose will be 70 Gray(Gy) at 2Gy/fraction, 35 fractions, Monday to Friday, for 7 weeks.
  Starting on the first day of radiotherapy, patients will be treated with pembrolizumab 200 milligrams (mg) intravenous (IV) every 3 weeks for 6 doses.
- Week 20 Assessment - Pembrolizumab Concomitant With and Post 7 Weeks of Radiation: Week 20 Quality of life Measurements
  All patients will receive Intensity Modulated Radiotherapy Treatments (IMRT) as per standard of care. The total dose will be 70 Gray(Gy) at 2Gy/fraction, 35 fractions, Monday to Friday, for 7 weeks.
  Starting on the first day of radiotherapy, patients will be treated with pembrolizumab 200 milligrams (mg) intravenous (IV) every 3 weeks for 6 doses.
Arm/Group | Baseline Assessment - Pembrolizumab Concomitant With and Post 7 Weeks of Radiation | Week 10 Assessment - Pembrolizumab Concomitant With and Post 7 Weeks of Radiation | Week 20 Assessment - Pembrolizumab Concomitant With and Post 7 Weeks of Radiation
Number analyzed (Participants) | 26 | 26 | 26
score on a scale
  PWB | 23.26 [21.41 to 25.11] | 17.63 [14.94 to 20.32] | 19.81 [16.81 to 22.81]
  SFWB | 22.26 [20.02 to 24.5] | 21.54 [19.50 to 23.57] | 23.40 [21.33 to 25.46]
  EWB | 18.12 [16.52 to 19.72] | 17.85 [15.36 to 20.34] | 17.59 [15.64 to 19.55]
  FWB | 19.00 [16.29 to 21.71] | 14.04 [11.20 to 16.87] | 16.74 [13.80 to 19.68]
  HNC | 24.57 [22.38 to 26.75] | 14.75 [12.67 to 16.84] | 18.92 [16.29 to 21.55]

ADVERSE EVENTS:
Time Frame: From day 1 of treatment up to 40 weeks after the end of treatment
Arm/Group | Pembrolizumab Concomitant With and Post 7 Weeks of Radiation
All-Cause Mortality (participants affected / at risk) | 7/29
Serious Adverse Events (participants affected / at risk) | 6/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab Concomitant With and Post 7 Weeks of Radiation (N=29)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Weight loss (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab Concomitant With and Post 7 Weeks of Radiation (N=29)
Abdominal pain (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 4
Allergic reaction (Immune system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 13
Anorexia (Metabolism and nutrition disorders) | 5
Anxiety (Psychiatric disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Aspartate aminotransferase increased (Investigations) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1
Blood bilirubin increased (Investigations) | 8
Blurred vision (Eye disorders) | 2
Bronchial infection (Infections and infestations) | 1
Chills (General disorders) | 4
Constipation (Gastrointestinal disorders) | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Creatinine increased (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 4
Depression (Psychiatric disorders) | 2
Dermatitis radiation (Injury, poisoning and procedural complications) | 24
Diarrhea (Gastrointestinal disorders) | 5
Dizziness (Nervous system disorders) | 1
Dry mouth (Gastrointestinal disorders) | 24
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dysgeusia (Nervous system disorders) | 24
Dysphagia (Gastrointestinal disorders) | 11
Dysphasia (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 2
Edema limbs (General disorders) | 2
Eye disorders - Other, specify (Eye disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 19
Fever (General disorders) | 3
Flu like symptoms (General disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4
Headache (Nervous system disorders) | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 9
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypotension (Vascular disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Insomnia (Psychiatric disorders) | 4
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 2
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 5
Lymph node pain (Blood and lymphatic system disorders) | 1
Lymphedema (Vascular disorders) | 3
Lymphocyte count decreased (Investigations) | 26
Memory impairment (Nervous system disorders) | 1
Mucosal infection (Infections and infestations) | 7
Mucositis oral (Gastrointestinal disorders) | 24
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 16
Neck edema (General disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 2
Neutrophil count decreased (Investigations) | 3
Non-cardiac chest pain (General disorders) | 1
Oral pain (Gastrointestinal disorders) | 4
Pain (General disorders) | 4
Papulopustular rash (Infections and infestations) | 1
Paresthesia (Nervous system disorders) | 1
Platelet count decreased (Investigations) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Salivary gland infection (Infections and infestations) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 10
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Tooth infection (Infections and infestations) | 1
Tracheal hemorrhage (Injury, poisoning and procedural complications) | 1
Tremor (Nervous system disorders) | 2
Trismus (Musculoskeletal and connective tissue disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary retention (Renal and urinary disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Weight gain (Investigations) | 1
Weight loss (Investigations) | 25
White blood cell decreased (Investigations) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT02609503/Prot_SAP_000.pdf